CLINICAL TRIAL: NCT02766465
Title: A Study to Compare Bone Marrow Transplantation to Standard Care in Adolescents and Young Adults With Severe Sickle Cell Disease (BMT CTN 1503)
Brief Title: Bone Marrow Transplantation vs Standard of Care in Patients With Severe Sickle Cell Disease (BMT CTN 1503)
Acronym: STRIDE2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Blood and Marrow Transplant Clinical Trials Network (Network); Dana-Farber Cancer Institute (Other); National Marrow Donor Program (Other); Emory University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BMT CTN 1503; 1U01HL128568-01 (NIH)
Record Dates: First submitted 2016-05-06; First posted 2016-05-09 (Estimated); Results first posted 2024-09-24 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Sickle Cell Disease
Keywords: Sickle Cell Disease; Young Adults; Phase II Trial; Hematopoietic Cell Transplantation (HCT); Human Leukocyte Antigen (HLA)
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — Busulfan; fludarabine; fludarabine phosphate; thymoglobulin; Bone Marrow Transplantation; Hematocrit; Tacrolimus; Methotrexate; Standard of Care; Alemtuzumab; Whole-Body Irradiation; Sirolimus; Melphalan; Granulocyte Colony-Stimulating Factor

STUDY DESIGN:
Intervention Model Description: Patients are enrolled without a known donor. All patients have 180 days from confirmation of eligibility to confirm a donor. Patients with a donor will be assigned to the Donor Arm and receive HCT; patients without a donor will be assigned to the no donor arm and continue receiving standard of care for their SCD.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Donor Arm (Experimental): Donor Arm patients will undergo hematopoietic cell transplant. Patients with a matched unrelated donor will receive a bone marrow transplant (unless PBSC graft is pre-approved per section 2.5.1 using a preparative regimen with Busulfan, Fludarabine and rabbit ATG. Patients with an HLA-identical sibling donor can receive a transplant using one of three regimens:
  A. Busulfan, Fludarabine, and rabbit ATG using a bone marrow graft (preferred regimen) B. Alemtuzumab/TBI 300 cGy using a peripheral blood graft C. Alemtuzumab, fludarabine, melphalan using a bone marrow graft
  Interventions: Drug: Busulfan; Drug: Fludarabine; Drug: r-ATG; Procedure: Hematopoietic Cell Transplant; Drug: Tacrolimus; Drug: Methotrexate; Drug: Alemtuzumab; Drug: Total Body Irradiation (TBI); Drug: Sirolimus; Drug: Melphalan; Drug: G-CSF
- No-Donor Arm (Active Comparator): No-donor arm patients will continue with standard of care per their SCD physician.
  Interventions: Procedure: Standard of Care

INTERVENTIONS:
Drug: Busulfan — A:
  Busulfan dose will be 3.2 mg/kg administered as a single daily dose IV on days -8 through -5 with dosing adjusted using targeted pharmacokinetics.
  Other Names: Busulfex
  Arms: Donor Arm
Drug: Fludarabine — A:
  Fludarabine dose will be 35 mg/m^2/day administered IV on days -7 through -3 (total fludarabine dose is 175 mg/m^2).
  C:
  Fludarabine 30mg/m2 IV dose will be given on Days -8, -7, -6, -5, -4
  Other Names: Fludara
  Arms: Donor Arm
Drug: r-ATG — A:
  r-ATG will be administered IV on day -6 at 0.5mg/kg, on day -5 at 1 mg/kg and on days -4, -3 and -2 at 1.5mg/kg (total r-ATG dose is 6 mg/kg).
  Other Names: Rabbit antithymocyte globulin
  Arms: Donor Arm
Procedure: Hematopoietic Cell Transplant — A,B,C:
  Day 0 is the day of transplantation.
  Other Names: Bone Marrow Transplant; BMT; HCT
  Arms: Donor Arm
Drug: Tacrolimus — A:
  Tacrolimus commences on day -3 and extends through day +180 after transplantation with doses adjusted to maintain appropriate levels according to institutional guidelines.
  C:
  Tacrolimus at therapeutic doses through Day 180, then taper per institutional guidelines
  Other Names: Prograf®
  Arms: Donor Arm
Drug: Methotrexate — A:
  Methotrexate will be administered intravenously on day+1 at 15mg/m^2, day+3 at 10mg/m^2, day+6 at 10mg/m^2, and day+11 at 10mg/m^2.
  C:
  Methotrexate IV 7.5 mg/m2 dose will be given on Days +1, 3, +6 following transplant
  Other Names: MTX
  Arms: Donor Arm
Procedure: Standard of Care — Continue to receive standard of care treatment per patient's SCD physician.
  Arms: No-Donor Arm
Drug: Alemtuzumab — B:
  Alemtuzumab 0.03 mg/kg IV dose will be given on Day -7, Alemtuzumab 0.1 mg/kg IV dose will be given on Day -6, Alemtuzumab 0.3 mg/kg IV dose will be given on Day -5,-4,-3
  C:
  Alemtuzumab test dose 3 mg IV once 24 hours prior to 1st dose of Alemtuzumab Alemtuzumab 10 mg IV, 15 mg IV, 20 mg IV given on Days -22 through Day -18. Alemtuzumab doses may be administered between Days -22 and -18 but are required to be on three consecutive days.
  Other Names: Lemtrada
  Arms: Donor Arm
Drug: Total Body Irradiation (TBI) — Total Body Irradiation 300 cGY on Day -2
  Arms: Donor Arm
Drug: Sirolimus — Sirolimus at therapeutic doses through day 180, then taper per institutional guidelines if donor CD3+ >50%
  Other Names: Rapamune
  Arms: Donor Arm
Drug: Melphalan — C:
  Melphalan 140 mg/m2 IV dose will be given on Day -3
  Other Names: Alkeran
  Arms: Donor Arm
Drug: G-CSF — G-CSF 5 μg/kg/day continue until neutrophil engraftment.
  Other Names: Granulocyte colony-stimulating factor
  Arms: Donor Arm

SUMMARY:
This is a clinical trial that will compare survival and sickle related outcomes in adolescents and young adults with severe sickle cell disease after bone marrow transplantation and standard of care. The primary outcome is 2-year overall survival.

DETAILED DESCRIPTION:
This is a prospective phase II multi-center trial of hematopoietic stem cell transplantation or standard of care based on availability of HLA-matched related or unrelated donor after confirmation of clinical eligibility. In order to minimize bias assignment to either treatment arm, clinical eligibility to both treatment arms are similar and donor availability is not known at referral. HLA typing and donor search is initiated upon confirmation of clinical eligibility for the study. Additionally, all analyses of primary and secondary endpoints will follow the Intent-to-Treat principle to address potential bias introduced by participants with donors not proceeding to transplantation or those without a matched donor receiving transplantation with less well-matched donors.

The primary outcome is 2-year overall survival. Our hypothesis is that patients who receive bone marrow transplantation will experience early deaths but that this will plateau by 2 years after transplantation. Patients who receive standard of care will not experience early death but will succumb to their disease at a rate much higher than the general population. Therefore, the goal of the study is to establish that the difference in the proportion of patients surviving is not significantly more than 15% lower in the donor arm at 2-years after assignment to treatment arm.

Secondary endpoints will compare changes in sickle cell disease related events (pulmonary hypertension, cerebrovascular events, renal function, avascular necrosis, leg ulcer) and functional outcomes [6-minute walk distance (6MWD), health-related quality of life, cardiac function, pulmonary function, and mean pain intensity as assessed by a multidimensional electronic pain diary] from baseline to 2-years after assignment to treatment arms.

Additionally for patients assigned to the donor arm and expected to undergo transplantation, hematopoietic recovery, graft rejection, acute and chronic graft-versus-host disease, other significant transplant-related complications and disease-free survival will be reported.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 15 and < 41 years
2. Severe sickle cell disease [Hemoglobin SS (Hb SS), Hemoglobin SC (Hb SC) or Hemoglobin SBeta thalassemia (Hb Sβ) genotype] with at least 1 of the following manifestations (a-e):

   1. Clinically significant neurologic event (stroke) or any neurological deficit lasting > 24 hours;
   2. History of two or more episodes of acute chest syndrome (ACS) in the 2-year period preceding enrollment despite the institution of supportive care measures (i.e. asthma therapy);
   3. An average of three or more pain crises per year in the 2-year period preceding enrollment (required intravenous pain management in the outpatient or inpatient hospital setting). Clinical documentation of pain management in the inpatient or outpatient setting is required.
   4. Administration of regular RBC transfusion therapy, defined as receiving 8 or more transfusion events per year (in the 12 months before enrollment) to prevent vaso-occlusive clinical complications (i.e. pain, stroke, and acute chest syndrome)
   5. An echocardiographic finding of tricuspid valve regurgitant jet (TRJ) velocity ≥ 2.7 m/sec.
   6. Ongoing high impact chronic pain on a majority of days per month for ≥ 6 months as defined as ONE or more of the following: Chronic pain without contributory SCD complications, OR Mixed pain type in which chronic pain is occurring at site(s) (arms, back, chest, or abdominal pain) unrelated to any sites associated with Contributory SCD complications (e.g. leg ulcers and/or avascular necrosis).

   i. High impact chronic pain is identified as those reporting "severe interference" with life activities OR "usually or always" experiencing a limitation of their life or work activities including household chores. (See guidelines for identifying HICP in the BMT CTN 1503 Manual of Procedures) ii. Contributory SCD complications are defined as clinical signs (e.g. presence of leg ulcers) or clinical assessments (e.g. imaging confirmation of splenic infarct or avascular necrosis). Chronic pain attributed solely to contributory SCD complications is excluded.
3. Adequate physical function as measured by all of the following:

   1. Karnofsky/Lansky performance score ≥ 60
   2. Cardiac function: Left ventricular ejection fraction (LVEF) > 40%; or LV shortening fraction > 26% by cardiac echocardiogram or by Multi Gated Acquisition Scan (MUGA).
   3. Pulmonary function:

   a. Pulse oximetry with a baseline O2 saturation of ≥ 85% b. Diffusing capacity of the lung for carbon monoxide (DLCO) > 40% (corrected for hemoglobin) d. Renal function: Serum creatinine ≤ 1.5 x the upper limit of normal for age as per local laboratory and 24 hour urine creatinine clearance >70 mL/min; or GFR > 70 mL/min/1.73 m2 by radionuclide Glomerular Filtration Rate (GFR).

   e. Hepatic function:
   1. Serum conjugated (direct) bilirubin < 2x upper limit of normal for age as per local laboratory. Participants are not excluded if the serum conjugated (direct) bilirubin is >2x the upper limit of normal for age as per local laboratory and: There is evidence of a hyperhemolytic reaction after a recent RBC transfusion, OR there is evidence of moderate direct hyperbilirubinemia defined as direct serum bilirubin < 5 times ULN and not caused by underlying hepatic diseasePatients
   2. alanine aminotransferase (ALT) and aspartate aminotransferase (AST) < 5 times upper limit of normal as per local laboratory.

Additional inclusion required for donor arm participants to proceed with transplant

1. Liver MRI (≤ 90 days prior to initiation of transplant conditioning) to document hepatic iron content is required for participants who are currently receiving ≥8 packed red blood cell transfusions for ≥1 year or have received ≥20 packed red blood cell transfusions (cumulative). Participants who have hepatic iron content ≥7 mg Fe/ g liver dry weight by liver MRI must have a liver biopsy and histological examination/documentation of the absence of cirrhosis, bridging fibrosis and active hepatitis (≤ 90 days prior to initiation of transplant conditioning).
2. Lack of clinical or radiologic evidence of a recent neurologic event (such as stroke or transient ischemic attack) by Cerebral MRI/MRA within 30 days prior to initiating transplant conditioning. Subjects with clinical or radiologic evidence of a recent neurologic event will be deferred for ≥ 6 months with repeat cerebral MRI/MRA to ensure stabilization of the neurologic event prior to proceeding to transplantation
3. Documentation of participant's willingness to use approved contraception method until discontinuation of all immunosuppressive medications is to be documented in the medical record corresponding with the consent conference.

Exclusion Criteria:

1. HLA typing with a donor search prior to referral (consultation with HCT physician).

   1. If a subject has had HLA typing and a related donor search that did not identify a suitably matched relative (i.e., sibling) at any time, and also did not have an unrelated donor search, the patient will be considered eligible.
   2. If a subject has had HLA typing and a related donor search that did not identify a suitably matched relative (i.e., sibling) at any time and had an unrelated donor search that did not identify a suitably matched unrelated donor ≥ 1 year prior to enrollment, the patient will be considered eligible.
   3. If a subject has had HLA typing with no related donor search and had an unrelated donor search that did not identify a suitably matched unrelated donor ≥ 1 year prior to enrollment, the patient will be considered eligible.
   4. Subjects with a known HLA-identical sibling or HLA-matched unrelated donor are excluded
2. Uncontrolled bacterial, viral or fungal infection in the 6 weeks before enrollment.
3. Seropositivity for HIV.
4. Previous HCT or solid organ transplant.
5. Participation in a clinical trial in which the patient received an investigational drug or device must be discontinued at enrollment.
6. A history of substance abuse as defined by version IV of the Diagnostic & Statistical Manual of Mental Disorders (DSM IV).
7. Demonstrated lack of compliance with prior medical care as determined by referring physician.
8. Pregnant or breast feeding females.
9. Inability to receive HCT due to alloimmunization, defined as the inability to receive packed red blood cell (pRBC) transfusion therapy.

Ages: 15 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 138 (Actual)
Dates: Start 2017-03-16 (Actual); Primary Completion 2023-05-02 (Actual); Study Completion 2023-08-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary Eapen, MD, Study Director — Center for International Blood and Marrow Transplant Research
Locations (35):
- United States (35):
  - Benioff Children's Hospital at Oakland, Oakland, California
  - Children's National Medical Center, Washington D.C., District of Columbia
  - University of Florida Gainsville, Gainesville, Florida
  - Foundation for Sickle Cell Research/Florida Sickle Inc., Hollywood, Florida
  - University of Miami, Miami, Florida
  - Grady Memorial Hospital, Atlanta, Georgia
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - Emory University, Atlanta, Georgia
  - Augusta University Medical Center, Augusta, Georgia
  - University of Iowa, Iowa City, Iowa
  - Children's Hospital of New Orleans, New Orleans, Louisiana
  - Dana Farber Cancer Institute/Brigham & Women's Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute/Massachusetts General Hospital, Boston, Massachusetts
  - Boston University, Boston, Massachusetts
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Washington University/St. Louis Children's Hospital, St Louis, Missouri
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - New York Presbyterian Brooklyn Methodist Hospital, Brooklyn, New York
  - Cohen Children's Medical Center, New Hyde Park, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Weill Cornell Medical College, New York, New York
  - Montefiore Medical Center/Albert Einstein School of Medicine, The Bronx, New York
  - University of North Carolina Hospital at Chapel Hill, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Ohio State University, Columbus, Ohio
  - University of Oklahoma, Oklahoma City, Oklahoma
  - Oregon Health Sciences University, Portland, Oregon
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - University of Texas Health Sciences Center, Houston, Texas
  - Baylor College of Medicine/The Methodist Hospital, Houston, Texas
  - University of Texas/MD Anderson CRC, Houston, Texas
  - University of Virginia, Charlottesville, Virginia
  - Virginia Commonwealth University, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: Yes
Results will be published in a manuscript and supporting information submitted to NIH BioLINCC (including data dictionaries, case report forms, data submission documentation, documentation for outcomes dataset, etc where indicated).
Supporting Information: Study Protocol, ICF
Time Frame: Within 6 months of official study closure at participating sites.
Access Criteria: Available to the public
URL: https://biolincc.nhlbi.nih.gov/home/

REFERENCES:
- [Result] Walters MC, Eapen M, Liu Y, El Rassi F, Waller EK, Levine JE, Strouse JJ, Antin JH, Parikh SH, Bakshi N, Dampier C, Jaroscak JJ, Bergmann S, Wong T, Kota V, Pace B, Lekakis LJ, Lulla P, Nickel RS, Kasow KA, Popat U, Smith W, Yu L, DiFronzo N, Geller N, Kamani N, Klings ES, Hassell K, Mendizabal A, Sullivan K, Neuberg D, Krishnamurti L. Hematopoietic cell transplant compared with standard care in adolescents and young adults with sickle cell disease. Blood Adv. 2025 Mar 11;9(5):955-965. doi: 10.1182/bloodadvances.2024013926. PMID 39471440
- [Derived] Leonard A, Furstenau D, Abraham A, Darbari DS, Nickel RS, Limerick E, Fitzhugh C, Hsieh M, Tisdale JF. Reduction in vaso-occlusive events following stem cell transplantation in patients with sickle cell disease. Blood Adv. 2023 Jan 24;7(2):227-234. doi: 10.1182/bloodadvances.2022008137. PMID 36240296
- [Derived] Krishnamurti L, Neuberg DS, Sullivan KM, Kamani NR, Abraham A, Campigotto F, Zhang W, Dahdoul T, De Castro L, Parikh S, Bakshi N, Haight A, Hassell KL, Loving R, Rosenthal J, Smith SL, Smith W, Spearman M, Stevenson K, Wu CJ, Wiedl C, Waller EK, Walters MC. Bone marrow transplantation for adolescents and young adults with sickle cell disease: Results of a prospective multicenter pilot study. Am J Hematol. 2019 Apr;94(4):446-454. doi: 10.1002/ajh.25401. Epub 2019 Feb 11. PMID 30637784
- See also: Blood and Marrow Transplant Clinical Trials Network Website — https://bmtctn.net/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: BMT CTN 1503's enrollment was between March 2017 and August 2021. The study opened to accrual on March 16, 2017 with activated 37 centers. The study closed to accrual on August 31, 2021 and study completed on May 2, 2023. A total of 138 eligible participants were enrolled to Segment 0 from 31 centers.
Pre-assignment Details: Among 138 enrolled patients, 123 were biologically assigned and enrolled in Segment A. Of the 15 who were not biologically assigned, 2 died prior to assignment due to SCD complications, 10 withdrew consent, 2 lost to follow-up, and 1 was removed per physician decision. Of the 123 biologically assigned patients, 28 patients across 13 institutions were assigned to the Donor Arm and 95 patients across 26 institutions were assigned to the No Donor Arm. In the donor arm 24 patients were transplanted.
Period: Overall Study
Arm/Group | Donor Arm | No-Donor Arm
Started | 28 | 95
Completed | 28 | 85
Not Completed | 0 | 10
Not completed — Withdrawal by Subject | 0 | 10

BASELINE CHARACTERISTICS:
Population: The total number of participants who were biologically assigned and permitted the analysis of their data was 113. Of these 85 participants were assigned to the No Donor Arm and 28 were assigned to the Donor Arm. For Severity of SCD Criteria, participants reported represent patients with disease severity in the corresponding diseases as specified in the Measure Description.
Groups:
- Total: Total of all reporting groups
Arm/Group | Donor Arm | No-Donor Arm | Total
Number analyzed (Participants) | 28 | 85 | 113
Age, Continuous [Median (Full Range); unit: years] | 29.1 [15.6 to 40.8] | 25.9 [15.6 to 39.3] | 26.2 [15.6 to 40.8]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 39 | 54
  Male | 13 | 46 | 59
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 8 | 12
  Not Hispanic or Latino | 24 | 75 | 99
  Unknown or Not Reported | 0 | 2 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 1 | 5 | 6
  Black or African American | 26 | 73 | 99
  Other | 1 | 2 | 3
  Unknown | 0 | 3 | 3
  Not answered | 0 | 2 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African American | 12 | 41 | 53
  African Black (both parents African) | 0 | 7 | 7
  Black (NOS) | 13 | 22 | 35
  Caribbean Black | 1 | 2 | 3
  Middle Eastern | 0 | 1 | 1
  Puerto Rican | 1 | 1 | 2
  Saudi Arabian | 0 | 1 | 1
  South or Central American | 0 | 1 | 1
  South or Central American Black | 0 | 1 | 1
  White (NOS) | 1 | 3 | 4
  Not answered | 0 | 2 | 2
  Unknown | 0 | 3 | 3
Sickle Cell Disease Type [Count of Participants; unit: Participants] — Sickle cell disease is a group of inherited disorders in which hemoglobin, the protein found in the red blood cells that carry oxygen throughout the body, is mutated so that the cells can take on a sickled shape at low oxygen levels. The cells become rigid and can block blood flow to the rest of the body. Sickle cell disease types are designated by the types of mutations in hemoglobin. The most common type of sickle cell disease has two copies of hemoglobin S (HbSS), but other mutations such a C, beta thalassemia, or OArab can pair with S to yield HbSC, HbS beta thalassemia or HbS-OArab.
  Participants
    HbSS | 21 | 67 | 88
    HbSC | 1 | 4 | 5
    HbS beta thalassemia | 2 | 9 | 11
    HbS-OArab | 0 | 1 | 1
    Unknown | 4 | 4 | 8
Severity of SCD Criteria [Count of Participants; unit: Participants] — Patients can report multiple criteria. Disease severity per an Eligibility Review Committee by >=1 of the following criteria: clinically significant neurologic event (stroke) or neurological deficit lasting >24 hrs; >=2 episodes of acute chest syndrome in the 2 years preceding enrollment; >=6 pain crises in the 2 years preceding enrollment requiring intravenous pain management; >=8 red blood cell transfusion events in the 12 months preceding enrollment; tricuspid valve regurgitant jet velocity >=2.7 m/sec; ongoing high impact chronic pain on a majority of days per month for >=6 months.
  Participants
    Neurologic | 7 | 7 | 14
    Acute Chest Syndrome (ACS) | 1 | 14 | 15
    Pain Crises | 17 | 62 | 79
    Red Blood Cell (RBC) Transfusion | 7 | 13 | 20
    Tricuspid valve Regurgitant Jet Velocity (TRJV) | 1 | 9 | 10
    High Impact Chronic Pain | 10 | 19 | 29

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Overall Survival (OS) at 2 Years After Biologic Assignment
Description: Due to incomplete accrual, there was not adequate statistical power to analyze the primary endpoint as specified. Instead, point estimates for the observed proportion of patients surviving at two years post-biologic assignment in each arm were generated descriptively, with 95% CI, using the Kaplan Meier methodology. The event of interest was death from any cause.
Time Frame: 2 Years
Population: Using the intent-to-treat principle, participants remained in their assigned treatment arm regardless of treatment received.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Donor Arm | No-Donor Arm
Number analyzed (Participants) | 28 | 85
percentage of participants | 89 [78 to 100] | 94 [87 to 99]

2. Secondary Outcome: Frequencies of Sickle Cell Disease (SCD) Events of Special Interest
Description: Examination of the occurrence of the SCD-related events was performed. Participants can have multiple events. The following sickle cell disease related events of special interest (SCD-EOSI) are expected events for all participants, regardless of biologic assignment:
  * pulmonary hypertension
  * significant cerebrovascular events, including: stroke; transient ischemic attack; seizure
  * renal function compromise, including: proteinuria; increased creatinine grades ≥2 per CTCAE version 4.0
  * avascular necrosis of the hip or shoulder
  * leg ulcers
  * acute chest syndrome (ACS) requiring hospitalization
  * vaso-occlusive pain crisis (VOC) requiring hospitalization or administration of parenteral opioid drugs in an outpatient setting. Self-reported events without clinical documentation should not be included.
Time Frame: 2 Years
Population: as for outcome 1
Measure: Number; unit: event
Arm/Group | Donor Arm | No-Donor Arm
Number analyzed (Participants) | 28 | 85
event
  Pulmonary hypertension at 1 yr | 1 | 6
  Significant cerebrovascular event including stroke, transient ischemic attack, and seizure at 1 yr | 8 | 4
  Renal function compromise at 1 yr | 7 | 14
  Avascular necrosis at 1 yr | 4 | 11
  Leg ulceration at 1 yr | 1 | 4
  Acute chest syndrome with hospitalization at 1 yr | 3 | 18
  Vaso-occlusive pain w/ hospitalization or parenteral opioid drugs in outpatient setting at 1 yr | 11 | 161
  Any event leading to an advanced care setting or intensive care unit admission/transfer at 1 yr | 5 | 5
  Pulmonary hypertension at 2 yrs | 1 | 7
  Significant cerebrovascular event including stroke, transient ischemic attack, and seizure at 2 yrs | 1 | 6
  Renal function compromise at 2 yrs | 4 | 8
  Avascular necrosis at 2 yrs | 1 | 8
  Leg ulceration at 2 yrs | 0 | 1
  Acute chest syndrome with hospitalization at 2 yrs | 0 | 10
  Vaso-occlusive pain w/ hospitalization or parenteral opioid drugs in outpatient setting at 2 yrs | 3 | 144
  Any event leading to an advanced care setting or intensive care unit admission/transfer at 2 yrs | 1 | 6
Statistical Analysis 1: Comparison: Donor Arm vs No-Donor Arm; This is the result comparing severe vaso-occlusive pain (VOC) with hospitalization or parenteral opioid drugs in outpatient setting between two biologically assigned arms during the first year after biologic assignment. The null hypothesis is that there is no difference in biologically assigned arms during the first year after assignment; Test type: Superiority; p < 0.001, Wilcoxon (Mann-Whitney) — Statistical significance was determined using a pre-specified threshold of 0.05
Statistical Analysis 2: Comparison: Donor Arm vs No-Donor Arm; This is the result comparing significant cerebrovascular event between two biologically assigned arms during the first year after biologic assignment. Significant cerebrovascular event includes stroke, transient ischemic attack, and seizure. The null hypothesis is that there is no difference in biologically assigned arms during the first year after assignment; Test type: Superiority; p = 0.027, Wilcoxon (Mann-Whitney) — Statistical significance was determined using a pre-specified threshold of 0.05
Statistical Analysis 3: Comparison: Donor Arm vs No-Donor Arm; This is the result comparing severe Vaso-occlusive pain (VOC) with hospitalization or parenteral opioid drugs in outpatient setting between two biologically assigned arms during the second year after biologic assignment. The null hypothesis is that there is no difference in biologically assigned arms during the second year after assignment; Test type: Superiority; p < 0.001, Wilcoxon (Mann-Whitney) — Statistical significance was determined using a pre-specified threshold of 0.05

3. Secondary Outcome: Change in 6-minute Walk Distance (6MWD) Assessment From Baseline
Description: The 6-minute walk distance (6MWD) test is a test to measure how far you can walk in 6 minutes. It is used in this study to assess exercise capacity. The number of meters that a participant could walk in 6 minutes was selected as a direct measurement of physical function.
Time Frame: Baseline, 2 years
Population: Participants that are biologically assigned to different arms and that completed both the baseline and 2-year assessment; this follows the intent-to-treat principle.
Measure: Median (Full Range); unit: meter
Arm/Group | Donor Arm | No-Donor Arm
Number analyzed (Participants) | 7 | 32
meter | -71 [-175 to 161] | -26 [-374 to 343]
Statistical Analysis 1: Comparison: Donor Arm vs No-Donor Arm; This is the result comparing 6MWD from 2 years after biologic assignment to baseline between two biologically assigned arms. The null hypothesis is that there is no difference between biologically assigned arms; Test type: Superiority; p = 0.869, Wilcoxon (Mann-Whitney) — Statistical significance was determined using a pre-specified threshold of 0.05

4. Secondary Outcome: Change in Transcuspid Regurgitant Jet Velocity (TRJV) Assessment From Baseline
Description: Transcuspid regurgitant jet velocity (TRJV) is a measure of how fast blood is pumped through one of the heart valves on the right side of the heart, measured using an ultrasound of the heart (echocardiogram). Higher values can indicate pulmonary hypertension and more severe sickle cell disease. Increasing TRJV over time indicates worsening disease.
Time Frame: Baseline, 2 years
Population: as for outcome 3
Measure: Median (Full Range); unit: meters per second (m/s)
Arm/Group | Donor Arm | No-Donor Arm
Number analyzed (Participants) | 4 | 16
meters per second (m/s) | 0.1 [-0.7 to 0.9] | 0.05 [-3.1 to 2.5]
Statistical Analysis 1: Comparison: Donor Arm vs No-Donor Arm; This is the result comparing TRJV from 2 years after biologic assignment to baseline between two biologically assigned arms. The null hypothesis is that there is no difference between biologically assigned arms; Test type: Superiority; p = 0.636, Wilcoxon (Mann-Whitney) — Statistical significance was determined using a pre-specified threshold of 0.05

5. Secondary Outcome: Change in Albuminuria Assessment From Baseline
Description: Albuminuria is the ratio of albumin (a protein) in the urine to creatinine in the urine. This may be assessed based on a 24-hour urine sample or a spot urine sample. Albumin in the urine may indicate kidney disease. Increases in albuminuria over time indicate increasing renal (kidney) disease.
Time Frame: Baseline, 2 years
Population: as for outcome 3
Measure: Median (Full Range); unit: mg of albumin per gram of creatine
Arm/Group | Donor Arm | No-Donor Arm
Number analyzed (Participants) | 0 | 6
mg of albumin per gram of creatine |  | 0 [-9 to 98]

6. Secondary Outcome: Health-Related Quality of Life (HRQoL) Component Physical Function Changes From Baseline
Description: Health-Related Quality of Life (HRQoL) assessed using the NIH's PROMIS 57 instrument. Physical Function asks about degree of difficulty in performing activities of daily living such as housework, errands, and going up and down stairs. It is scored from 0 to 10 and converted to a standardized T-score with mean 50 and standard deviation 10. A higher T-score represents better physical function.
Time Frame: Baseline, 2 years
Population: as for outcome 3
Measure: Median (Full Range); unit: T-score
Arm/Group | Donor Arm | No-Donor Arm
Number analyzed (Participants) | 10 | 37
T-score | 5 [-10 to 16] | 1 [-20 to 26]
Statistical Analysis 1: Comparison: Donor Arm vs No-Donor Arm; This is the result comparing Physical Function changes from 2 years after biologic assignment to baseline between two biologically assigned arms. The null hypothesis is that there is no difference between biologically assigned arms; Test type: Superiority; p = 0.242, Wilcoxon (Mann-Whitney) — Statistical significance was determined using a pre-specified threshold of 0.05

7. Secondary Outcome: Health-Related Quality of Life (HRQoL) Component Anxiety Changes From Baseline
Description: Health-Related Quality of Life (HRQoL) assessed using the NIH's PROMIS 57 instrument. Anxiety asks about the frequency of feelings of fear, worry, and anxiety. It is scored from 0 to 10 and converted to a standardized T-score with mean 50 and standard deviation 10. A higher T-score represents more anxiety.
Time Frame: Baseline, 2 years
Population: as for outcome 3
Measure: Median (Full Range); unit: T-score
Arm/Group | Donor Arm | No-Donor Arm
Number analyzed (Participants) | 9 | 37
T-score | 0 [-21 to 4] | 0 [-13 to 20]
Statistical Analysis 1: Comparison: Donor Arm vs No-Donor Arm; This is the result comparing Anxiety changes from 2 years after biologic assignment to baseline between two biologically assigned arms. The null hypothesis is that there is no difference between biologically assigned arms; Test type: Superiority; p = 0.343, Wilcoxon (Mann-Whitney) — Statistical significance was determined using a pre-specified threshold of 0.05

8. Secondary Outcome: Health-Related Quality of Life (HRQoL) Component Depression Changes From Baseline
Description: Health-Related Quality of Life (HRQoL) assessed using the NIH's PROMIS 57 instrument. Depression asks about the frequency of feelings of worthlessness, failure, unhappiness and depression. It is scored from 0 to 10 and converted to a standardized T-score with mean 50 and standard deviation 10. A higher T-score represents more depression.
Time Frame: Baseline, 2 years
Population: as for outcome 3
Measure: Median (Full Range); unit: T-score
Arm/Group | Donor Arm | No-Donor Arm
Number analyzed (Participants) | 9 | 37
T-score | 0 [-10 to 8] | 0 [-20 to 26]
Statistical Analysis 1: Comparison: Donor Arm vs No-Donor Arm; This is the result comparing Depression changes from 2 years after biologic assignment to baseline between two biologically assigned arms. The null hypothesis is that there is no difference between biologically assigned arms; Test type: Superiority; p = 0.491, Wilcoxon (Mann-Whitney) — Statistical significance was determined using a pre-specified threshold of 0.05

9. Secondary Outcome: Health-Related Quality of Life (HRQoL) Component Fatigue Score Changes in From Baseline
Description: Health-Related Quality of Life (HRQoL) assessed using the NIH's PROMIS 57 instrument. Fatigue asks about the extent to which fatigue interferes with physical functioning and completing tasks. It is scored from 0 to 10 and converted to a standardized T-score with mean 50 and standard deviation 10. A higher T-score represents more fatigue.
Time Frame: Baseline, 2 years
Population: as for outcome 3
Measure: Median (Full Range); unit: T-score
Arm/Group | Donor Arm | No-Donor Arm
Number analyzed (Participants) | 10 | 37
T-score | -13 [-28 to 1] | 0 [-22 to 20]
Statistical Analysis 1: Comparison: Donor Arm vs No-Donor Arm; This is the result comparing fatigue score changes from 2 years after biologic assignment to baseline between two biologically assigned arms. The null hypothesis is that there is no difference between biologically assigned arms; Test type: Superiority; p = 0.003, Wilcoxon (Mann-Whitney) — Statistical significance was determined using a pre-specified threshold of 0.05

10. Secondary Outcome: Health-Related Quality of Life (HRQoL) Component Sleep Disturbance Changes From Baseline
Description: Health-Related Quality of Life (HRQoL) assessed using the NIH's PROMIS 57 instrument. Sleep Disturbance asks about the quality of sleep and the frequency with which sleep was restless or difficult to achieve. It is scored from 0 to 10 and converted to a standardized T-score with mean 50 and standard deviation 10. A higher T-score represents more sleep disturbance.
Time Frame: Baseline, 2 years
Population: as for outcome 3
Measure: Median (Full Range); unit: T-score
Arm/Group | Donor Arm | No-Donor Arm
Number analyzed (Participants) | 10 | 37
T-score | 1 [-17 to 15] | 0 [-24 to 14]
Statistical Analysis 1: Comparison: Donor Arm vs No-Donor Arm; This is the result comparing Sleep Disturbance changes from 2 years after biologic assignment to baseline between two biologically assigned arms. The null hypothesis is that there is no difference between biologically assigned arms; Test type: Superiority; p = 0.594, Wilcoxon (Mann-Whitney) — Statistical significance was determined using a pre-specified threshold of 0.05

11. Secondary Outcome: Health-Related Quality of Life (HRQoL) Component Participation in Social Roles Score Changes From Baseline
Description: Health-Related Quality of Life (HRQoL) assessed using the NIH's PROMIS 57 instrument. Participation in Social Roles asks about the frequency of limitations of social activities with friends and family. It is scored from 0 to 10 and converted to a standardized T-score with mean 50 and standard deviation 10. A higher T-score represents more satisfaction with participation in social roles.
Time Frame: Baseline, 2 years
Population: as for outcome 3
Measure: Median (Full Range); unit: T-score
Arm/Group | Donor Arm | No-Donor Arm
Number analyzed (Participants) | 10 | 36
T-score | 15 [-4 to 22] | 2 [-25 to 21]
Statistical Analysis 1: Comparison: Donor Arm vs No-Donor Arm; This is the result comparing social roles score changes from 2 years after biologic assignment to baseline between two biologically assigned arms. The null hypothesis is that there is no difference between biologically assigned arms; Test type: Superiority; p = 0.003, Wilcoxon (Mann-Whitney) — Statistical significance was determined using a pre-specified threshold of 0.05

12. Secondary Outcome: Health-Related Quality of Life (HRQoL) Component Pain Interference Score Changes From Baseline
Description: Health-Related Quality of Life (HRQoL) assessed using the NIH's PROMIS 57 instrument. Pain Interference asks about the frequency with which pain interferes with household chores, social activities and enjoyment of life. It is scored from 0 to 10 and converted to a standardized T-score with mean 50 and standard deviation 10. A higher T-score represents more pain interference in daily life.
Time Frame: Baseline, 2 years
Population: as for outcome 3
Measure: Median (Full Range); unit: T-score
Arm/Group | Donor Arm | No-Donor Arm
Number analyzed (Participants) | 10 | 37
T-score | -12 [-21 to 16] | -1 [-26 to 22]
Statistical Analysis 1: Comparison: Donor Arm vs No-Donor Arm; This is the result comparing pain interference score changes from 2 years after biologic assignment to baseline between two biologically assigned arms. The null hypothesis is that there is no difference between biologically assigned arms; Test type: Superiority; p = 0.071, Wilcoxon (Mann-Whitney) — Statistical significance was determined using a pre-specified threshold of 0.05

13. Secondary Outcome: Health-Related Quality of Life (HRQoL) Component Pain Intensity Changes From Baseline
Description: Health-Related Quality of Life (HRQoL) assessed using the NIH's PROMIS 57 instrument. Pain Intensity is scored from 0 to 10 reflecting the level of pain over the previous 7 days. A score of 0 reflects no pain; a score of 10 reflects the maximum intensity of pain.
Time Frame: Baseline, 2 years
Population: as for outcome 3
Measure: Median (Full Range); unit: T-score
Arm/Group | Donor Arm | No-Donor Arm
Number analyzed (Participants) | 10 | 37
T-score | -0.5 [-5 to 2] | 0 [-6 to 9]
Statistical Analysis 1: Comparison: Donor Arm vs No-Donor Arm; This is the result comparing Pain Intensity changes from 2 years after biologic assignment to baseline between two biologically assigned arms. The null hypothesis is that there is no difference between biologically assigned arms; Test type: Superiority; p = 0.146, Wilcoxon (Mann-Whitney) — Statistical significance was determined using a pre-specified threshold of 0.05

14. Secondary Outcome: Health-Related Quality of Life (HRQoL) Component 28-Day Pain Diary Average Pain Intensity Changes From Baseline
Description: Health-Related Quality of Life (HRQoL) assessed using the NIH's PROMIS 57 instrument. The 28-Day Pain Diary Average Pain Intensity assesses pain on a score of 0 to 10 twice each day for 28 days. A score of 0 reflects no pain, and a score of 10 reflects maximum intensity of pain. The scores on a given day are averaged (if only one score is obtained on a given day, that score is taken as the measure), and then daily scores are averaged over the number of days on which a score is available.
Time Frame: Baseline, 2 years
Population: as for outcome 3
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Donor Arm | No-Donor Arm
Number analyzed (Participants) | 5 | 17
units on a scale | -0.08 [-4.28 to 1.24] | -0.25 [-2.89 to 1.75]
Statistical Analysis 1: Comparison: Donor Arm vs No-Donor Arm; This is the result comparing 28-Day Pain Diary Average Pain Intensity changes from 2 years after biologic assignment to baseline between two biologically assigned arms. The null hypothesis is that there is no difference between biologically assigned arms; Test type: Superiority; p = 0.649, Wilcoxon (Mann-Whitney) — Statistical significance was determined using a pre-specified threshold of 0.05

15. Secondary Outcome: Health-Related Quality of Life (HRQoL) Component ASCQ-Me Stiffness Changes From Baseline
Description: Health-Related Quality of Life (HRQoL) assessed using the NIH's PROMIS 57 instrument. The ASCQ-Me Stiffness Scale asks about the frequency and severity of joint stiffness. It is scored from 0 to 10 and converted to a standardized T-score with mean 50 and standard deviation 10. A higher T-score represents more stiffness.
Time Frame: Baseline, 2 years
Population: as for outcome 3
Measure: Median (Full Range); unit: T-score
Arm/Group | Donor Arm | No-Donor Arm
Number analyzed (Participants) | 10 | 37
T-score | -1 [-23 to 13] | 1 [-13 to 19]
Statistical Analysis 1: Comparison: Donor Arm vs No-Donor Arm; This is the result comparing ASCQ-Me Stiffness changes from 2 years after biologic assignment to baseline between two biologically assigned arms. The null hypothesis is that there is no difference between biologically assigned arms; Test type: Superiority; p = 0.207, Wilcoxon (Mann-Whitney) — Statistical significance was determined using a pre-specified threshold of 0.05

16. Secondary Outcome: Change in Pulmonary Function of Forced Expiratory Volume 1 Second (FEV1) From Baseline
Description: Pulmonary function is assessed by the change from baseline in Forced Expiratory Volume 1 second (FEV1). The complete pulmonary function test will include forced expiratory volume in 1 second (FEV1), forced vital capacity (FVC), ratio of FEV1 to FVC (FEV1/FVC), vital capacity (VC), total lung capacity (TLC), residual volume (RV), expiratory reserve volume (ERV), inspiratory capacity (IC), functional residual capacity (FRC), diffusing capacity for carbon monoxide (DLCO), and oxygen saturation.
Time Frame: Baseline, 2 years
Population: Analysis population includes participants that are biologically assigned to different arms and completed both baseline and 2-year assessment.
Measure: Median (Full Range); unit: percentage of FEV1
Arm/Group | Donor Arm | No-Donor Arm
Number analyzed (Participants) | 12 | 31
percentage of FEV1 | 2.5 [-20 to 14] | 0.0 [-87 to 21]
Statistical Analysis 1: Comparison: Donor Arm vs No-Donor Arm; This is the result comparing FEV1 changes from 2 years after biologic assignment to baseline between two biologically assigned arms. The null hypothesis is that there is no difference between biologically assigned arms; Test type: Superiority; p = 0.596, Wilcoxon (Mann-Whitney) — Statistical significance was determined using a pre-specified threshold of 0.05

17. Secondary Outcome: Change in Pulmonary Function of Forced Vital Capacity (FVC) From Baseline
Description: Pulmonary function is assessed by the change from baseline in forced vital capacity (FVC). The complete pulmonary function test will include forced expiratory volume in 1 second (FEV1), forced vital capacity (FVC), ratio of FEV1 to FVC (FEV1/FVC), vital capacity (VC), total lung capacity (TLC), residual volume (RV), expiratory reserve volume (ERV), inspiratory capacity (IC), functional residual capacity (FRC), diffusing capacity for carbon monoxide (DLCO), and oxygen saturation.
Time Frame: Baseline, 2 years
Population: as for outcome 16
Measure: Median (Full Range); unit: percentage of FVC
Arm/Group | Donor Arm | No-Donor Arm
Number analyzed (Participants) | 12 | 31
percentage of FVC | 1.5 [-23 to 10] | 0.0 [-15 to 25]
Statistical Analysis 1: Comparison: Donor Arm vs No-Donor Arm; This is the result comparing FVC changes from 2 years after biologic assignment to baseline between two biologically assigned arms. The null hypothesis is that there is no difference between biologically assigned arms; Test type: Superiority; p = 0.684, Wilcoxon (Mann-Whitney) — Statistical significance was determined using a pre-specified threshold of 0.05

18. Secondary Outcome: Change in Pulmonary Function of Ratio of FEV1 to FVC (FEV1/FVC) From Baseline
Description: Pulmonary function is assessed by the change from baseline in ratio of FEV1 to FVC (FEV1/FVC). The complete pulmonary function test will include forced expiratory volume in 1 second (FEV1), forced vital capacity (FVC), ratio of FEV1 to FVC (FEV1/FVC), vital capacity (VC), total lung capacity (TLC), residual volume (RV), expiratory reserve volume (ERV), inspiratory capacity (IC), functional residual capacity (FRC), diffusing capacity for carbon monoxide (DLCO), and oxygen saturation.
Time Frame: Baseline, 2 years
Population: as for outcome 16
Measure: Median (Full Range); unit: percentage of FEV1/FVC
Arm/Group | Donor Arm | No-Donor Arm
Number analyzed (Participants) | 10 | 30
percentage of FEV1/FVC | 0.5 [-8 to 28] | 0.5 [-97 to 21]
Statistical Analysis 1: Comparison: Donor Arm vs No-Donor Arm; This is the result comparing FEV1/FVC changes from 2 years after biologic assignment to baseline between two biologically assigned arms. The null hypothesis is that there is no difference between biologically assigned arms; Test type: Superiority; p = 0.863, Wilcoxon (Mann-Whitney) — Statistical significance was determined using a pre-specified threshold of 0.05

19. Secondary Outcome: Change in Pulmonary Function of Vital Capacity (VC) From Baseline
Description: Pulmonary function is assessed by the change from baseline in vital capacity (VC). The complete pulmonary function test will include forced expiratory volume in 1 second (FEV1), forced vital capacity (FVC), ratio of FEV1 to FVC (FEV1/FVC), vital capacity (VC), total lung capacity (TLC), residual volume (RV), expiratory reserve volume (ERV), inspiratory capacity (IC), functional residual capacity (FRC), diffusing capacity for carbon monoxide (DLCO), and oxygen saturation.
Time Frame: Baseline, 2 years
Population: as for outcome 16
Measure: Median (Full Range); unit: percentage of VC
Arm/Group | Donor Arm | No-Donor Arm
Number analyzed (Participants) | 6 | 13
percentage of VC | 0.5 [-26 to 13] | 2 [-14 to 23]
Statistical Analysis 1: Comparison: Donor Arm vs No-Donor Arm; This is the result comparing VC changes from 2 years after biologic assignment to baseline between two biologically assigned arms. The null hypothesis is that there is no difference between biologically assigned arms; Test type: Superiority; p = 0.455, Wilcoxon (Mann-Whitney) — Statistical significance was determined using a pre-specified threshold of 0.05

20. Secondary Outcome: Change in Pulmonary Function of Total Lung Capacity (TLC) From Baseline
Description: Pulmonary function is assessed by the change from baseline in total lung capacity (TLC). The complete pulmonary function test will include forced expiratory volume in 1 second (FEV1), forced vital capacity (FVC), ratio of FEV1 to FVC (FEV1/FVC), vital capacity (VC), total lung capacity (TLC), residual volume (RV), expiratory reserve volume (ERV), inspiratory capacity (IC), functional residual capacity (FRC), diffusing capacity for carbon monoxide (DLCO), and oxygen saturation.
Time Frame: Baseline, 2 years
Population: as for outcome 16
Measure: Median (Full Range); unit: percentage of TLC
Arm/Group | Donor Arm | No-Donor Arm
Number analyzed (Participants) | 6 | 23
percentage of TLC | -1.0 [-23 to 7] | 0 [-10 to 86]
Statistical Analysis 1: Comparison: Donor Arm vs No-Donor Arm; This is the result comparing TLC changes from 2 years after biologic assignment to baseline between two biologically assigned arms. The null hypothesis is that there is no difference between biologically assigned arms; Test type: Superiority; p = 0.767, Wilcoxon (Mann-Whitney) — Statistical significance was determined using a pre-specified threshold of 0.05

21. Secondary Outcome: Change in Pulmonary Function of Residual Volume (RV) From Baseline
Description: Pulmonary function is assessed by the change from baseline in residual volume (RV). The complete pulmonary function test will include forced expiratory volume in 1 second (FEV1), forced vital capacity (FVC), ratio of FEV1 to FVC (FEV1/FVC), vital capacity (VC), total lung capacity (TLC), residual volume (RV), expiratory reserve volume (ERV), inspiratory capacity (IC), functional residual capacity (FRC), diffusing capacity for carbon monoxide (DLCO), and oxygen saturation.
Time Frame: Baseline, 2 years
Population: as for outcome 16
Measure: Median (Full Range); unit: percentage of RV
Arm/Group | Donor Arm | No-Donor Arm
Number analyzed (Participants) | 5 | 21
percentage of RV | 6 [-27 to 36] | -11 [-95 to 49]
Statistical Analysis 1: Comparison: Donor Arm vs No-Donor Arm; This is the result comparing RV changes from 2 years after biologic assignment to baseline between two biologically assigned arms. The null hypothesis is that there is no difference between biologically assigned arms; Test type: Superiority; p = 0.241, Wilcoxon (Mann-Whitney) — Statistical significance was determined using a pre-specified threshold of 0.05

22. Secondary Outcome: Change in Pulmonary Function of Expiratory Reserve Volume (ERV) From Baseline
Description: Pulmonary function is assessed by the change from baseline in expiratory reserve volume (ERV). The complete pulmonary function test will include forced expiratory volume in 1 second (FEV1), forced vital capacity (FVC), ratio of FEV1 to FVC (FEV1/FVC), vital capacity (VC), total lung capacity (TLC), residual volume (RV), expiratory reserve volume (ERV), inspiratory capacity (IC), functional residual capacity (FRC), diffusing capacity for carbon monoxide (DLCO), and oxygen saturation.
Time Frame: Baseline, 2 years
Population: as for outcome 16
Measure: Median (Full Range); unit: percentage of ERV
Arm/Group | Donor Arm | No-Donor Arm
Number analyzed (Participants) | 6 | 21
percentage of ERV | 9.5 [-5 to 36] | -2 [-47 to 61]
Statistical Analysis 1: Comparison: Donor Arm vs No-Donor Arm; This is the result comparing ERV changes from 2 years after biologic assignment to baseline between two biologically assigned arms. The null hypothesis is that there is no difference between biologically assigned arms; Test type: Superiority; p = 0.268, Wilcoxon (Mann-Whitney) — Statistical significance was determined using a pre-specified threshold of 0.05

23. Secondary Outcome: Change in Pulmonary Function of Inspiratory Capacity (IC) From Baseline
Description: Pulmonary function is assessed by the change from baseline in inspiratory capacity (IC). The complete pulmonary function test will include forced expiratory volume in 1 second (FEV1), forced vital capacity (FVC), ratio of FEV1 to FVC (FEV1/FVC), vital capacity (VC), total lung capacity (TLC), residual volume (RV), expiratory reserve volume (ERV), inspiratory capacity (IC), functional residual capacity (FRC), diffusing capacity for carbon monoxide (DLCO), and oxygen saturation.
Time Frame: Baseline, 2 years
Population: as for outcome 16
Measure: Median (Full Range); unit: percentage of IC
Arm/Group | Donor Arm | No-Donor Arm
Number analyzed (Participants) | 3 | 18
percentage of IC | -1 [-15 to 13] | -4.5 [-20 to 22]
Statistical Analysis 1: Comparison: Donor Arm vs No-Donor Arm; This is the result comparing IC changes from 2 years after biologic assignment to baseline between two biologically assigned arms. The null hypothesis is that there is no difference between biologically assigned arms; Test type: Superiority; p > 0.999, Wilcoxon (Mann-Whitney) — Statistical significance was determined using a pre-specified threshold of 0.05

24. Secondary Outcome: Change in Pulmonary Function of Functional Residual Capacity (FRC) From Baseline
Description: Pulmonary function is assessed by the change from baseline in functional residual capacity (FRC). The complete pulmonary function test will include forced expiratory volume in 1 second (FEV1), forced vital capacity (FVC), ratio of FEV1 to FVC (FEV1/FVC), vital capacity (VC), total lung capacity (TLC), residual volume (RV), expiratory reserve volume (ERV), inspiratory capacity (IC), functional residual capacity (FRC), diffusing capacity for carbon monoxide (DLCO), and oxygen saturation.
Time Frame: Baseline, 2 years
Population: as for outcome 16
Measure: Median (Full Range); unit: percentage of FRC
Arm/Group | Donor Arm | No-Donor Arm
Number analyzed (Participants) | 4 | 10
percentage of FRC | 3 [-8 to 12] | -3.5 [-28 to 40]
Statistical Analysis 1: Comparison: Donor Arm vs No-Donor Arm; This is the result comparing FRC changes from 2 years after biologic assignment to baseline between two biologically assigned arms. The null hypothesis is that there is no difference between biologically assigned arms; Test type: Superiority; p = 0.832, Wilcoxon (Mann-Whitney) — Statistical significance was determined using a pre-specified threshold of 0.05

25. Secondary Outcome: Change in Pulmonary Function of Diffusing Capacity for Carbon Monoxide (DLCO) From Baseline
Description: Pulmonary function is assessed by the change from baseline in diffusing capacity for carbon monoxide (DLCO). The complete pulmonary function test will include forced expiratory volume in 1 second (FEV1), forced vital capacity (FVC), ratio of FEV1 to FVC (FEV1/FVC), vital capacity (VC), total lung capacity (TLC), residual volume (RV), expiratory reserve volume (ERV), inspiratory capacity (IC), functional residual capacity (FRC), diffusing capacity for carbon monoxide (DLCO), and oxygen saturation.
Time Frame: Baseline, 2 years
Population: as for outcome 16
Measure: Median (Full Range); unit: percentage of DLCO
Arm/Group | Donor Arm | No-Donor Arm
Number analyzed (Participants) | 10 | 28
percentage of DLCO | -4 [-22 to 43] | 0 [-40 to 62]
Statistical Analysis 1: Comparison: Donor Arm vs No-Donor Arm; This is the result comparing DLCO changes from 2 years after biologic assignment to baseline between two biologically assigned arms. The null hypothesis is that there is no difference between biologically assigned arms; Test type: Superiority; p = 0.370, Wilcoxon (Mann-Whitney) — Statistical significance was determined using a pre-specified threshold of 0.05

26. Secondary Outcome: Change in Pulmonary Function of Oxygen Saturation From Baseline
Description: Pulmonary function is assessed by the change from baseline in oxygen saturation. The complete pulmonary function test will include forced expiratory volume in 1 second (FEV1), forced vital capacity (FVC), ratio of FEV1 to FVC (FEV1/FVC), vital capacity (VC), total lung capacity (TLC), residual volume (RV), expiratory reserve volume (ERV), inspiratory capacity (IC), functional residual capacity (FRC), diffusing capacity for carbon monoxide (DLCO), and oxygen saturation.
Time Frame: Baseline, 2 years
Population: as for outcome 16
Measure: Median (Full Range); unit: percentage of oxygen saturation
Arm/Group | Donor Arm | No-Donor Arm
Number analyzed (Participants) | 11 | 33
percentage of oxygen saturation | 1 [-2 to 6] | 0 [-3 to 6]
Statistical Analysis 1: Comparison: Donor Arm vs No-Donor Arm; This is the result comparing oxygen saturation changes from 2 years after biologic assignment to baseline between two biologically assigned arms. The null hypothesis is that there is no difference between biologically assigned arms; Test type: Superiority; p = 0.094, Wilcoxon (Mann-Whitney) — Statistical significance was determined using a pre-specified threshold of 0.05;

27. Secondary Outcome: Frequencies of Infections
Description: All Grade 2 and 3 infections were reported according to the BMT CTN Technical Manual of Procedures (MOP) after biological assignment. The frequency of Grade 2-3 infections are tabulated by biological assignment at the event level.
Time Frame: 2 years
Population: as for outcome 1
Measure: Number; unit: infection
Arm/Group | Donor Arm | No-Donor Arm
Number analyzed (Participants) | 28 | 85
infection
  Herpes Zoster | 2 | 0
  Clostridium difficile | 4 | 2
  Human Herpes Virus - 6 | 2 | 0
  Staphylococcus (coag +) | 1 | 0
  Respiratory Syncytial virus | 1 | 0
  Other Bacteria | 2 | 0
  Rhinovirus | 2 | 0
  Streptococcus | 1 | 0
  Other Viral | 5 | 2
  Epstein-Barr Virus | 3 | 0
  Staphylococcus (NOS) | 2 | 0
  Staphylococcus (coag -) | 2 | 1
  Escherichia coli | 3 | 1
  Cytomegalovirus | 2 | 0
  Influenza | 1 | 0
  Klebsiella | 0 | 1
  Pseudomonas | 0 | 1
  Bacillus | 0 | 1
  Enterococcus | 0 | 1
  Gram Negative Rod (NOS) | 0 | 1
  Staphylococcus | 0 | 1

28. Secondary Outcome: Percentage of Participants With Grades II-IV Acute GVHD at Day 180 After Biological Assignment
Description: The time interval from day 0 of transplant until grade II-IV aGVHD will be described for each treatment arm using the the cumulative incidence estimator developed by Gray, with death prior to aGVHD treated as a competing risk. Estimates and 95% CIs of the cumulative incidence of grade II-IV aGVHD will be provided at Day 180 after day 0 of transplant and compared between matched related and matched unrelated donors using the Gray test.
  Acute GVHD was graded according to the BMT CTN Technical Manual of Operating Procedures (MOP). Higher aGVHD grade indicate worse outcomes. Grade I is defined as Skin stage 1-2 and stage 0 for both GI and liver. Grade II is stage 3 skin, stage 1 GI, or stage 1 liver. Grade III is stage 2-3 GI or stage 2-3 liver. Grade IV is stage 4 skin or stage 4 liver.
Time Frame: 180 days after biological assignment
Population: Patients who enrolled on the donor arm and received transplant
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- HLA Matched Sibling Donor: For patients who enrolled on the donor arm, 10 patients received transplant from sibling donors.
- Unrelated Donor: For patients who enrolled on the donor arm, 14 patients received transplant from unrelated donors.
Arm/Group | HLA Matched Sibling Donor | Unrelated Donor
Number analyzed (Participants) | 10 | 14
percentage of participants | 30 [6.2 to 59] | 46 [18 to 71]
Statistical Analysis 1: Comparison: HLA Matched Sibling Donor vs Unrelated Donor; The null hypothesis is that there is no difference of grade II-IV acute GVHD in patients who received different donor type at transplant; Test type: Superiority; p = 0.313, Gray's test for cumulative Incidence — Statistical significance was determined using a pre-specified threshold of 0.05

29. Secondary Outcome: Percentage of Participants With Chronic GVHD at Day 600 After Biological Assignment
Description: Chronic GVHD was collected according to the recommendations of the NIH Consensus Conference. Eight organs will be scored on a 0-3 scale to reflect degree of chronic GVHD involvement. Liver and pulmonary function test results and use of systemic therapy for treatment of chronic GVHD was also recorded. Percentage of Participants with chronic GVHD (cGVHD) at Day 600 was estimated with 95% confidence intervals for each donor type group using the cumulative incidence estimate, treating death prior to cGVHD as a competing event.
Time Frame: Day 600 after biological assignment
Population: Patients who enrolled on the donor arm and received transplant.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- HLA-matched Sibling Donor: For patients who enrolled on the donor arm, 10 patients received transplant from sibling donors.
Arm/Group | HLA-matched Sibling Donor | Unrelated Donor
Number analyzed (Participants) | 10 | 14
percentage of participants | 30 [6.2 to 59] | 57 [26 to 79]
Statistical Analysis 1: Comparison: HLA-matched Sibling Donor vs Unrelated Donor; The null hypothesis is that there is no difference of chronic GVHD in patients who received different donor type at transplant; Test type: Superiority; p = 0.233, Gray's test for cumulative Incidence — Statistical significance was determined using a pre-specified threshold of 0.05

30. Secondary Outcome: Number of Participants With Primary and Secondary Graft Failure
Description: Primary graft failure defined as never achieving ANC ≥ 500/µL or never achieving ≥ 5% donor whole blood or myeloid chimerism (myeloid is preferable) assessed by bone marrow or peripheral blood chimerism assays by day +42 post-transplant. Second infusion of hematopoietic cells is also considered indicative of primary graft failure by day +42 post-transplant. Secondary graft failure is defined as < 5% donor whole blood or myeloid chimerism (myeloid is preferable) in peripheral blood or bone marrow beyond day +42 post-transplant in patients with prior documentation of hematopoietic recovery with ≥ 5% donor cells by day +42 post-transplant. Second infusion of hematopoietic cells is also considered indicative of secondary graft failure.
Time Frame: 2 years
Population: Analysis population includes transplanted participants who were biologically assigned to donor arm.
Measure: Number; unit: participants
Arm/Group | Donor Arm
Number analyzed (Participants) | 24
participants
  Primary graft failure | 0
  Secondary graft failure | 3

ADVERSE EVENTS:
Time Frame: Adverse event reporting requirements become effective at the time of the participant's biologic assignment, and up to 2 years
Description: AE reporting was conducted according to the BMT CTN's Manual of Operating Procedures. Unexpected, serious AEs (SAEs) were reported through an expedited AE reporting system. Expected AEs were reported using National Cancer Institute (NCI)'s Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0 at regular intervals.
Arm/Group | Donor Arm | No-Donor Arm
All-Cause Mortality (participants affected / at risk) | 3/28 | 5/85
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/85
Other Adverse Events (participants affected / at risk) | 14/28 | 65/85
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Donor Arm (N=28) | No-Donor Arm (N=85)
PRES (Nervous system disorders) | 1 (1) | 0 (0)
ACCIDENTAL DRUG OVERDOSE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
TONIC CLONIC SEIZURE (Nervous system disorders) | 1 (1) | 0 (0)
EPILEPTIC SEIZURES (Nervous system disorders) | 1 (1) | 0 (0)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
SICKLE CELL CRISIS AND BIPAP (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
DEATH (General disorders) | 0 (0) | 2 (2)
ACUTE SUBARACHNOID HEMORRHAGE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
ACUTE RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
GRADE 4 MUCOSITIS ORAL (Gastrointestinal disorders) | 1 (1) | 0 (0)
MULTIPLE ORGAN FAILURE (General disorders) | 1 (1) | 0 (0)
HYPERTENSION MANAGEMENT (Vascular disorders) | 1 (1) | 0 (0)
POSTERIOR REVERSIBLE ENCEPHALOPATHY (Nervous system disorders) | 2 (3) | 0 (0)
ACUTE CHEST SYNDROME (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
SEPSIS (Infections and infestations) | 1 (1) | 1 (1)
MUCOSITIS (General disorders) | 1 (1) | 0 (0)
HYPERGLYCEMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
CARDIAC ARRES (Cardiac disorders) | 0 (0) | 1 (1)
ACUTE PYELONEPHRITIS (Infections and infestations) | 1 (2) | 0 (0)
CONGESTIVE HEART FAILURE (Cardiac disorders) | 0 (0) | 1 (1)
END STAGE RENAL DISEASE (Renal and urinary disorders) | 0 (0) | 1 (1)
SEPTIC SHOCK (Infections and infestations) | 1 (1) | 0 (0)
GRAFT VERSUS HOST DISEASE (Immune system disorders) | 1 (1) | 0 (0)
ACUTE CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 0 (0) | 1 (1)
RESPIRATORY DISTRES (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (7) — During the second year following biologic assignment
Significant cerebrovascular event (Nervous system disorders) | 1 (1) | 5 (6) — During the second year following biologic assignment
Renal function compromise (Renal and urinary disorders) | 3 (4) | 6 (8) — During the second year following biologic assignment
Avascular necrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 6 (8) — During the second year following biologic assignment
Leg ulceration (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — During the second year following biologic assignment
Acute chest syndrome with hospitalization (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 8 (10) — During the second year following biologic assignment
Vaso-occlusive pain with hospitalization or parenteral opioid drugs in outpatient setting (Blood and lymphatic system disorders) | 2 (3) | 59 (144) — During the second year following biologic assignment
Bacterial, Fungal, and Viral Infections (Infections and infestations) | 14 (33) | 10 (12)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (6) — During the first year following biologic assignment
Significant cerebrovascular event (Nervous system disorders) | 5 (8) | 3 (4) — During the first year following biologic assignment
Renal function compromise (Renal and urinary disorders) | 5 (7) | 11 (14) — During the first year following biologic assignment
Avascular necrosis (Musculoskeletal and connective tissue disorders) | 4 (4) | 10 (11) — During the first year following biologic assignment
Leg ulceration (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (4) — During the first year following biologic assignment
Acute chest syndrome with hospitalization (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 12 (18) — During the first year following biologic assignment
Vaso-occlusive pain with hospitalization or parenteral opioid drugs in outpatient setting (Blood and lymphatic system disorders) | 10 (11) | 65 (161) — During the first year following biologic assignment

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2023-06-08): https://cdn.clinicaltrials.gov/large-docs/65/NCT02766465/Prot_SAP_ICF_001.pdf